CLINICAL TRIAL: NCT01272557
Title: Sorafenib Plus Doxorubicin Versus Sorafenib Alone for the Treatment of Advanced Hepatocellular Carcinoma: a Randomized Phase II Trial
Acronym: SoraDox
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PD Dr. med. Matthias Dollinger (Other)
Responsible Party: Sponsor-Investigator, PD Dr. med. Matthias Dollinger, PD. Dr. med., Martin-Luther-Universität Halle-Wittenberg
Organization: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SoraDox
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Liver Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib 400 mg bid (oral) continuously (Active Comparator): Sorafenib 400 mg bid (oral) continuously until progression or unacceptable toxicity).
  Interventions: Drug: Sorafenib
- q22d: Doxorubicin 60 mg/m2 i.v d1, Sorafenib 400 mg bid d3-19 (Experimental): During trial therapy period in Arm-A treated patients will receive doxorubicin infusion with 60mg/m² on day 1 every 21 days for maximum of 18 weeks (or 6 cycles) until a maximal dose of 360mg/m² are reached. Sorafenib 400mg bid (oral) will be administered from day 3-19 every 21 days during the trial therapy period
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 60 mg/m2 i.v. on day 1 every 21 days Sorafenib 400 mg bid (oral) from day 3-19 every 21 days. Maximum accumulative dose of doxorubicin: 360 mg/m2 (thereafter sorafenib monotherapy continuously until progression or unacceptable toxicity).
  Arms: q22d: Doxorubicin 60 mg/m2 i.v d1, Sorafenib 400 mg bid d3-19
Drug: Sorafenib — Sorafenib 400 mg bid (oral) continuously
  Arms: Sorafenib 400 mg bid (oral) continuously

SUMMARY:
This study is a prospective, randomized, open-label, multicenter phase IIB trial in order to determine time to progression of the combination therapy sorafenib plus doxorubicin against standard-of-care sorafenib in advanced HCC not amenable to non-systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-resectable locally advanced or metastasized HCC
* Subjects must have at least one tumor lesion that meets both of the following criteria:
* the lesion can be accurately measured in at least one dimension according to RECIST 1.1
* the lesion has not been previously treated with local therapy (such as surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation)
* Subjects who have received local therapy (such as surgery, radiation therapy, hepatic arterial therapy, chemoembolization, radiofrequency ablation, percutaneous ethanol injection or cryoablation) are eligible, provided that they have a target lesion which has not been subjected to local therapy. Local therapy must be completed at least 4 weeks prior to the baseline scan.
* Confirmation of disease by histology
* Liver function: Child Pugh stage A/B (5-7 points) only
* Tumor stage: BCLC stage C (or better)
* ECOG performance status 0-2
* Life expectancy of at least 12 weeks
* Age ≥ 18 years
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening and within 4 weeks before start of treatment:
* Hemoglobin ≥ 9.0 g/dl
* Absolute neutrophil count (ANC) ≥1.500/mm3
* Platelet count ≥ 70.000/μl
* Total bilirubin ≤ 3 mg/dl
* ALT and AST ≤ 5 x upper limit of normal
* Alkaline phosphatase < 4 x upper limit of normal
* PT-INR/PTT < 1.5 x upper limit of normal [Patients who are being therapeutically anticoagulated with an agent such as warfarin, phenprocoumon or heparin will NOT be allowed to participate]
* Serum creatinine ≤ 1.5 x upper limit of normal
* Signed and dated informed consent before start of any study specific procedure

Exclusion Criteria:

* Patients eligible for resection or transplantation
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study. However cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis and T1) or any cancer curatively treated > 3 years prior to entry is permitted
* Serious myocardial dysfunction: defined as absolute left ventricular ejection fraction (LVEF) < 50%, instable coronaropathy (MI more than 6 mo prior to study entry is allowed), cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted)
* Inadequately controlled hepatic complications (varices, encephalopathy)
* Untreated active Hepatitis B including HBs-Ag carriers; patients should be started on (prophylactic) anti-viral medication even without current viral replication
* Concomitant therapy with interferon (e.g. Hepatitis B/C) during study phase
* Uncontrolled arterial hypertension with systolic blood pressure >160 mmHg or diastolic blood pressure > 90 mm Hg despite optimal treatment
* Known history of HIV infection
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0)
* Symptomatic metastatic brain or meningeal tumors (unless the patient is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry)
* Patients with seizure disorder requiring medication (such as steroids or anti-epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Thrombotic or embolic events within the last 6 months
* Serious non-healing wound, fracture, or ulcer
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Women enrolled in this trial must use adequate barrier birth control measures during the course of the trial for at least 6 months after last administration of doxorubicin and 2 months after the last administration of sorafenib.
* Severe concomitant disease or psychiatric disorders
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known severe hypersensitivity to sorafenib, doxorubicin or any of the excipients
* Patients unable to swallow oral medications
* Incompliance / contraindications against study medication

Excluded therapies and medications, previous and concomitant:

* Previous systemic therapy for HCC
* Anticancer chemotherapy or immunotherapy or targeted therapy (except study medication) during the study or within 4 weeks of study entry.
* Radiotherapy during study or within 3 weeks of start of study drug. (Palliative radiotherapy will be allowed). Major surgery within 4 weeks of start of study
* Autologous bone marrow transplant or stem cell rescue within 4 months of study
* Use of biologic response modifiers, such as G-CSF, within 3 week of study entry. [G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction.] [Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 2 months prior to the study or during the study]
* Patients receiving anticoagulation therapy or ASS >100 mg/d
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry
* Prior exposure to the study drug.
* Any St. John's wort containing remedy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) according to RECIST 1.1 criteria | The follow-up period ends 12 months after enrolment of the last patient (end of study visit of the last patient unless he died earlier

SECONDARY OUTCOMES:
• Assessment of overall survival (OS) of disease control rate (CR, PR, SD) to RECIST 1.1 criteria and to EASL criteria • Assessment of safety and quality of life (FACT-Hep) and potential of biomarkers to predict the tumor response | The follow-up period ends 12 months after enrolment of the last patient (end of study visit of the last patient unless he died earlier).

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Medizinische Klinik und Poliklinik, Heinrich-Heine-Universität, Düsseldorf
  - Martin-Luther-University Halle-Wittenberg, Halle
  - Universitätsklinikum des Saarlande, Homburg/Saar
  - Ortenau Klinikum Lahr-Ettenheim, Lahr
  - Universitätsklinikum Leipzig, Leipzig
  - Klinikum Ludwigsburg, Ludwigsburg